CLINICAL TRIAL: NCT00074555
Title: Consortium for the Longitudinal Evaluation of African Americans With Early Rheumatoid Arthritis (CLEAR)
Brief Title: Registry for African Americans With Early Rheumatoid Arthritis
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: N01 AR02247; NIAMS-106
Record Dates: First submitted 2003-12-16; First posted 2003-12-17 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
Keywords: African American, Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand the causes of rheumatoid arthritis (RA), particularly in African Americans.

DETAILED DESCRIPTION:
RA is an autoimmune disease in which the body's immune system attacks its own tissues. It occurs in all races and ethnic groups and affects about two to three times as many women as men. Variations in certain genes that play a role in the immune system are associated with a tendency to develop RA. Some individuals without these genetic variations may develop this disease, while others who possess the variations never develop RA. Scientists believe that some environmental factors may play a part in triggering the disease process in people whose genetic makeup makes them susceptible to RA. This registry of African Americans with early RA will provide clinical and x-ray data and DNA to help scientists analyze genetic and nongenetic factors that might predict disease course and outcomes of RA in this population.

Participants in this registry will be enrolled in the study until they reach 5 years in their disease duration. For example, if a participant enters the study after 1 year of having RA, he or she will continue for 4 years. Participants will have three office visits (screening, 3 years' disease duration, and 5 years' disease duration) at which they will complete questionnaires and have blood samples taken, x-rays of their hands and feet, and DEXA scans. Between office visits, the study coordinator will call participants every 6 months to update any changes in medications or health problems.

ELIGIBILITY:
Inclusion Criteria

* African American
* Rheumatoid arthritis for less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African Americans
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2001-01; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Radiographic severity of rheumatoid arthritis in African Americans | 5 yr disease duration
  Initially seen at 5 yr disease duration. Later, became a cross-sectional (1 time visit).

CONTACTS AND LOCATIONS:
Overall Officials: S. Louis Bridges, Jr., MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Emory University, Atlanta, Georgia
  - Washington University at St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina